CLINICAL TRIAL: NCT00832143
Title: Effect of Referral Card on Neonatal Medical Care Seeking for Institutional Births in Urban Lucknow
Acronym: Referral Card
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King George's Medical University (Other)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Prof Shally Awasthi, Chattrapati Shahuji Maharaj Medical University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 819/R.Cell 04; ICMR 5/7/94/04/RHN
Record Dates: First submitted 2009-01-28; First posted 2009-01-29 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Neonatal Morbidity; Neonatal Illnesses
Keywords: neonatal illness; qualified care seeking; Behaviour change; Urban slums; India; Neonatal morbidity; Care seeking for neonatal illnesses; Qualified medical care seeking; Integrated management of neonatal and childhood illnesses (IMNCI)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Usual Care
- 2 (Experimental): Referral Card with one-to-one counseling
  Interventions: Behavioral: Referral Card with one-to-one counseling

INTERVENTIONS:
Behavioral: Referral Card with one-to-one counseling — A Referral Card (Neonatal Well-Being Card) along with one-to-one counseling to mothers within 48 hours of institutional delivery
  Arms: 2

SUMMARY:
Neonatal mortality rate in Uttar Pradesh, Northern India is 53.6 per thousand, and accounts for 8% of global neonatal deaths.It has been argued that prompt and appropriate care-seeking for sick neonates can substantially reduce neonatal mortality. This pre and post intervention trial was done to assess the impact of a pictorial "Neonatal referral Card" and one-to-one counseling of mothers on the qualified medical care-seeking behavior for sick neonates in urban Lucknow.

The study hypothesis was that the counseling on danger signs along with neonatal referral card has no impact on availing services of a qualified medical practitioner by caregivers of sick neonates.

DETAILED DESCRIPTION:
The study was conducted in two government maternity hospitals in Lucknow. Neonates enrolled in the pre intervention phase were followed up for 6 weeks+15 days but did not recieve the study intervention. While, the mothers of the neonates enrolled in the post intervention phase recieved the study intervention within 48 hours of institutional delivery.Enrollment and follow-up procedures were same in both the phases.

ELIGIBILITY:
Inclusion Criteria:

* Neonates born in the participating hospital within last 48 hours and the parents on which gave written informed consent to participate in the study.

Exclusion Criteria:

* Neonates presenting with any clinically detectable congenital malformation at birth or who required any resuscitation at birth or who were admitted for any morbidity immediately after birth or those who were not the residents of Lucknow or were likely to leave the city limits within next one month.

Max Age: 4 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1020 (Actual)
Dates: Start 2007-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
The utilization of health services of qualified medical care provider (attendance; hospitalization) for neonatal sickness | In neonatal period

SECONDARY OUTCOMES:
To assess the causes of failure of health seeking behavior for neonatal illnesses of the community | in neonatal period

CONTACTS AND LOCATIONS:
Locations (1):
- King George's Medical University, Lucknow, Uttar Pradesh, India

REFERENCES:
- [Result] Awasthi S, Srivastava NM, Pant S. Symptom-specific care-seeking behavior for sick neonates among urban poor in Lucknow, Northern India. J Perinatol. 2008 Dec;28 Suppl 2:S69-75. doi: 10.1038/jp.2008.169. PMID 19057571